CLINICAL TRIAL: NCT04587219
Title: An Open Study of the Safety, Tolerability and Immunogenicity of the "Gam-COVID-Vac"Vaccine Against COVID-19 (Solution for Intramuscular Injection) With the Participation of Volunteers in the Age Group Over 60 Years
Brief Title: The Study of "Gam-COVID-Vac" Vaccine Against COVID-19 With the Participation of Volunteers of 60 y.o and Older
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 05-Gam-COVID-Vac-2020
Record Dates: First submitted 2020-10-13; First posted 2020-10-14 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-10

CONDITIONS: Coronavirus Infection
Keywords: COVID-19; vaccine; vector vaccine; Immunologic Factors; SARS-CoV-2
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Gam-COVID-Vac vaccine

STUDY DESIGN:
Intervention Model Description: Open prospective non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gam COVID Vac Vaccine (Experimental): the test drug will be administered according to the prime-boost scheme: the introduction of component 1 (Ad26) will be carried out on the 1st day, and component 2(Ad5)- on the 21st day of the study.
  Interventions: Biological: Gam-COVID-Vac

INTERVENTIONS:
Biological: Gam-COVID-Vac — combined vector vaccine, 0,5ml/dose+0,5 ml/dose prime-boost immunization in days 1 (component I rAd26-S) and 21(component II rAd5-S)

SUMMARY:
The purpose of this study: to assess the safety, tolerability and immunogenicity of the drug "Gam-COVID-Vac", a solution for intramuscular injection, at various times after vaccination in volunteers over 60 years of age

DETAILED DESCRIPTION:
An open-ended prospective non-randomized study involving volunteers over the age of 60.

The study will include 110 volunteers. who will receive the test drug according to the prime-boost scheme: the introduction of component 1 will be carried out on the 1st day, and component 2 - on the 21st day of the study. Outpatient monitoring will be performed during 4 visits: on the 7th, 14th, 28th, and 42nd days after the vaccine administration Also two visits will be performed in the phone contact mode for 90 and 180 days

ELIGIBILITY:
Inclusion Criteria:

1. The written informed consent of the subject for participation in the study;
2. Men and women over the age of 60 years inclusive;
3. Negative result of research on HIV, hepatitis, syphilis;
4. negative test result for the presence of IgM and IgG antibodies to SARS CoV2 by enzyme immunoassay;
5. negative test result for COVID-2019, determined by PCR at the screening session;
6. The absence of a history COVID-2019;
7. No contact of the study subject with COVID-2019 patients for at least 14 days prior to inclusion in the study (according to the study participant);
8. Consent to use effective methods of contraception during the entire period of participation in the study;
9. A negative test for the presence of narcotic and psychoactive agents in urine at the screening visit;
10. A negative test for alcohol at screening visit;
11. negative pregnancy test (performed for women with preserved reproductive potential)
12. No history of severe postvaccinal reactions or postvaccinal complications after the use of immunobiological drugs;
13. absence of acute infectious and/or respiratory diseases for at least 14 days prior to inclusion in the study.

Exclusion Criteria:

1. any vaccination/immunization performed within 30 days prior to inclusion in The study;
2. therapy with steroids (with the exception of hormonal contraceptives and drugs used as hormone replacement therapy for menopause) and/or immunoglobulins or other blood products that did not end 30 days before inclusion in the study;
3. Therapy immunosuppressive drugs, which ended less than 3 months before inclusion in the study;
4. Subjects of the female gender during pregnancy or breastfeeding;
5. Postponed less than one year before inclusion in the study, acute coronary syndrome or stroke;
6. Tuberculosis, chronic systemic infections;
7. burdened allergic history (the presence in the history of information about anaphylactic shock, Quincke's edema, polymorphic exudative eczema, atopy, serum sickness), hypersensitivity or allergic reactions to the introduction of immunobiological drugs, known allergic reactions to the components of the drug, exacerbation of allergic diseases on the day of inclusion in the study;
8. the presence of a history of neoplasms (ICD codes C00-D09);
9. donation of blood or plasma (450 ml or more) less than 2 months before inclusion in the study;
10. Splenectomy in history;
11. Neutropenia (decrease in the absolute number of neutrophils less than 1000/mm3), agranulocytosis, significant blood loss, severe anemia (hemoglobin less than 80 g/l), a history of immunodeficiency for 6 months before inclusion in the study;
12. Subjects with an active form of the disease caused by the human immunodeficiency virus, syphilis, hepatitis B and C;
13. Anorexia, protein deficiency of any origin;
14. extensive tattoos at the sites of drug administration (deltoid muscle area), which do not allow to assess the local response to the introduction of ILP;
15. Alcoholism and drug addiction in history;
16. Consists on the account at the psychiatrist;
17. subject's participation in any other interventional clinical trial within 90 days prior to the start of this study;
18. any other condition of the research subject that, in the opinion of the research doctor, may prevent the completion of the study in accordance with The Protocol;
19. staff of research centers and other employees directly involved in the research (members of the research team) and their families.
20. severe comorbid diseases that, in the opinion of the research doctor, may prevent participation in the study.

    -

Ages: 60 Years to 111 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Changing of antibody levels against the SARS-CoV-2 glycoprotein S in 42 days | at days 0, 21, 28, 42
  Determination of antibody levels against the SARS-CoV-2 glycoprotein S measured by an ELISA vs. baseline values
Number of Participants With Adverse Events | through the whole study, an average of 180 days
  Determination of Number of Participants With Adverse Events

SECONDARY OUTCOMES:
Changing of of virus neutralizing antibody titer | at days 0, 28, 42
  Determination of virus neutralizing antibody titer
Changing of antigen-specific cellular immunity level | Time Frame: at days 0,28
  Determination of antigen-specific cellular immunity

CONTACTS AND LOCATIONS:
Overall Officials: Nikita Lomakin, MD, PhD, Principal Investigator — Federal state budgetary institution "Central clinical hospital with polyclinic" Of the office Of the President of the Russian Federation
Locations (1):
- Federal state budgetary institution "Central clinical hospital with polyclinic" Of the office Of the President of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No